CLINICAL TRIAL: NCT02387346
Title: The Contribution of the Cerebello-thalamo-cortical Circuit to the Pathology of Non-dopaminergic Responsive Parkinson's Disease Symptoms
Brief Title: The Cerebellum as a Potential Treatment Site for PD Motor Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Life Financial Movement Disorders Research and Rehabilitation Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4247
Record Dates: First submitted 2015-03-03; First posted 2015-03-13 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Real Stimulation (Experimental): Participants in this group will receive Repetitive Transcranial Magnetic Stimulation, characterized by 900 pulses at 1Hz over the medial cerebellum at 120% resting motor threshold of the right first dorsal interosseous.
  Interventions: Device: Magstim Rapid 2 Repetitive Transcranial Magnetic Stimulation
- Sham Stimulation (Sham Comparator): Participants will receive Sham Repetitive Transcranial Magnetic Stimulation by having the coil angled at 90 degrees to the scalp; this will allow adequate noise output from the stimulator in the absence on real magnetic stimulation.
  Interventions: Device: Magstim Rapid 2 Sham Stimulation

INTERVENTIONS:
Device: Magstim Rapid 2 Repetitive Transcranial Magnetic Stimulation
  Arms: Real Stimulation
Device: Magstim Rapid 2 Sham Stimulation
  Arms: Sham Stimulation

SUMMARY:
The role of the cerebello-thalamo-cortical loop in the generation of tremor, gait impairments and postural instability has been made evident. The current study will use a Magstim Rapid 2 to deliver rTMS with the aim of modulating the activity in the vermal/paravermal region of the cerebellum, and consequently the cerebello-thalamo-cortical pathway. Analysis of the effects of an acute session of stimulation will be made to determine the therapeutic potential of the protocol. Motor symptom improvement will be assessed immediately following stimulation to detect motor symptom improvement up to one hour following stimulation, providing insight into the effectiveness of the protocol to produce benefits which outlast the period of stimulation.

Participants will each receive one session of stimulation in the ON state of medication. A pre-assessment will be performed before beginning the session and a post-assessment will be performed immediately following stimulation. There will be two groups, which will both undergo the exact same protocol, however one group will receive real stimulation, and one group will receive sham stimulation.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with idiopathic Parkinson's disease
* ability to walk 10 metres unassisted
* ability to stand for 5 minutes unassisted
* understand verbal instructions in English

Exclusion Criteria:

* presence of brain implants (aneurysm clips, deep brain stimulation electrodes)
* cochlear implants
* diagnosed with vascular Parkinson's disease
* history or increased risk of seizure
* severe dyskinesia of neck muscles

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Gait (GaitRite carpet using Zeno software to measure spatial and temporal aspects of gait.) | Immediately post stimulation, effects up to one hour
  5 trials of self-paced gait on a GaitRite carpet using Zeno software to measure spatial and temporal aspects of gait.
Balance: Postural Stability Testing (quiet stance on a balance force plate) | Immediately post stimulation, effects up to one hour
  3 trials lasting 30 seconds each of quiet stance on a balance force plate, where postural deviations from a central reference point on the platform will give an overall measure of postural sway, as well as score in the medial-lateral and anterior-posterior direction
Balance: Sensory Integration Testing (modified clinical test of sensory integration on balance (m-CTSIB) | Immediately post stimulation, effects up to one hour
  In accordance with the modified clinical test of sensory integration on balance (m-CTSIB), where four trials lasting 20 seconds each measure balance during various sensory conditions: 1) eyes open, firm platform, 2) eyes closed, firm platform, 3) eyes open, foam platform, 4) eyes closed, foam platform.
Tremor: Kinesia Homeview Tablet (tremor magnitude, frequency and amplitude can be measured with wireless finger accelerometer) | Immediately post stimulation, effects up to one hour
  With the use of a wireless finger accelerometer, tremor magnitude, frequency and amplitude can be measured during the upper limb movement tasks (such as rapid alternation and pointing tasks)

CONTACTS AND LOCATIONS:
Overall Officials: Quincy J Almeida, PhD, Study Director — SunLife Financial Movement Disorders Research & Rehabilitation Centre, Wilfrid Laurier University
Locations (1):
- Sun Life Financial Movement Disorders Research & Rehabilitation Centre, Waterloo, Ontario, Canada